CLINICAL TRIAL: NCT04051437
Title: Therapeutic Plasma Exchange in Patients With Acute on Chronic Liver Failure: A Randomized Controlled Trial (PLEXAR)
Brief Title: Plasma Exchange in Acute on Chronic Liver Failure
Acronym: PLEXAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Dr. Pramod Kumar, Principal Investigator, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG/IEC34/07.2019-08
Record Dates: First submitted 2019-08-03; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Cirrhosis, Liver; Acute-On-Chronic Liver Failure
Keywords: Plasma exchange; Acute on chronic liver failure
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma exchange (Experimental): The consented patients will receive standard medical management with sessions of single volume plasma exchange with fresh frozen plasma and 5% human albumin.Plasma exchange session will be done on an alternate day to a maximum of 5 procedures.
  Interventions: Procedure: Plasma exchange
- Standard medical treatment (Active Comparator): The consented patients will receive standard medical treatment which includes adequate nutrition (35-45 Kcal/Kg with 1.5gm/Kg protein) diuretics, anti HE measures, appropriate antibiotics for infections, entecavir 0.5 mg once daily for hepatitis B, and steroids for autoimmune hepatitis.
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Procedure: Plasma exchange — During each plasma exchange session 3-4lt (1.2-1.3 times of plasma volume) of plasma will be exchanged with fresh frozen plasma and 5% albumin. Plasma exchange session will be done on an alternate day to a maximum of 5 procedures. PLEX will be discontinued if the patients Shows sustained clinical improvement, Receive liver transplantation, Refuses further PLEX session No improvement in clinical condition Intolerant to PLEX procedure
  Arms: Plasma exchange
Drug: Standard medical treatment — The consented patients will receive standard medical treatment which includes adequate nutrition (35-45 Kcal/Kg with 1.5gm/Kg protein) diuretics, anti HE measures, appropriate antibiotics for infections,tablet entecavir 0.5 mg once daily for hepatitis B, and steroids for autoimmune hepatitis.
  Arms: Standard medical treatment

SUMMARY:
Acute on chronic liver failure (ACLF) is a distinct syndrome in patients with chronic liver disease with rapid clinical deterioration and has high short term mortality within one month.Despite aggressive clinical care, only half of the patients could survive an episode of ACLF. The investigators hypothesized that the early treatment with therapeutic plasma exchange with plasma and albumin in ACLF patients might improve overall survival in carefully selected patients by removing cytokines, chemokines and toxic substances.

DETAILED DESCRIPTION:
Acute on chronic liver failure (ACLF) lacks a consensus definition and definitive management approaches. The various management strategies include treatment of acute insult, support of multiple organ systems and disease-specific medications such as antivirals for hepatitis B, steroids for alcoholic hepatitis, and autoimmune hepatitis. Despite aggressive clinical care, only half of the patients could survive an episode of ACLF. ACLF is a dynamic condition and has specific time-related disease course. Majority of patients of the patients attain their final grade of ACLF between 3 rd and 7th day and makes it an ideal time to assess the prognosis. Recently, liver transplantation option also explored in patients not responding to standard medical care and appeared promising. Early liver transplantation is considered if the baseline model for end-stage liver disease (MELD) score > 28, Asia pacific association for the study of the liver (APASL) ACLF Research Consortium (AARC) score of > 10, advanced hepatic encephalopathy in the absence of organ failures or overt sepsis. However, liver transplantation is feasible only in 25% cases and approximately 67% waitlist mortality. Treating ACLF patients early in the disease course, i.e., window period, may prevent multiorgan dysfunction and improve outcomes. Therefore, these alternative modalities can act as bridging to liver transplantation and hasten the spontaneous liver regeneration and hence, transplant-free recovery in some patients.

Plasma exchange has been shown to reduce cytokines, inflammatory mediators, and damage-associated molecular patterns. The early experience of therapeutic plasma exchange in patients with hepatitis B ACLF shows a survival benefit compared to standard of care. Changes in albumin quantity and quality are noted in patients with cirrhosis. An increase in oxidized albumin, ischemia-modified albumin, and albumin dimerization is observed ACLF patients and changes are more pronounced compared to cirrhotic patients. These changes are well correlated with short and long term mortality.

Hence the investigators hypothesized that the early treatment with therapeutic plasma exchange with plasma and albumin in ACLF patients improves overall survival in carefully selected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ACLF as per APASL criteria with AARC score of ≥8

Exclusion Criteria:

1. Uncontrolled sepsis
2. Septic shock requiring inotropes despite fluid resuscitation
3. Active or recent bleeding (unless controlled for >48 hours).
4. Severe thrombocytopenia (≤20×10^9/L)
5. Acute kidney injury with Creatinine > 2 or the need of RRT
6. Respiratory failure (Severe ARDS)
7. Chronic kidney disease
8. Hepatocellular carcinoma outside Milan criteria (1 nodule ≤5 cm or 3 nodules ≤3 cm)
9. HIV infection
10. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 90 days

SECONDARY OUTCOMES:
Transplant free survival | 90 days
Development of organ dysfunction | 28 days
Development of cirrhosis complications | 28 days
Improvement in Model for end stage liver disease score | 90 days

IPD SHARING:
Plan to Share IPD: No